CLINICAL TRIAL: NCT04614597
Title: A Study on Immunity Duration Against Polio Over 18 Months Infants After 2 or 3 Primary Doses Sabin Strain Inactivated Poliovirus Vaccine in China
Brief Title: A Study on Immunity Duration Against Polio Over 18 Months Infants After 2 or 3 Primary Doses Sabin IPV in China
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Collaborators: World Health Organization (Other); Shandong Province Centers for Disease Control and Prevention (Other)
Responsible Party: Principal Investigator, AN Zhijie, Researcher of National Immunization Program, Centers for Disease Control and Prevention, China
Other Study IDs: 201935
Record Dates: First submitted 2020-10-28; First posted 2020-11-04 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Poliomyelitis
Keywords: Inactivated Poliovirus Vaccine; Sabin strain
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Three-dose schedule for Sabin IPV: Subjects already vaccinated Sabin IPV at 2, 3, and 4 months of age, collected two blood samples and laboratory test results were available.
  Interventions: Biological: Sabin strain inactivated polio vaccine
- Two-dose schedule for Sabin IPV: Subjects already vaccinated Sabin IPV at 4 and 8-11 months of age, collected two blood samples and laboratory test results were available.
  Interventions: Biological: Sabin strain inactivated polio vaccine

INTERVENTIONS:
Biological: Sabin strain inactivated polio vaccine — Sabin IPVs have been given to participants in previously study, blood specimens will be collected once all the subjects reach the age of 18months.

SUMMARY:
In 2017, China CDC conducted a study titled "A Study of Immunogenicity and Seroconversion With Sabin IPV Schedules in China". At present, all the infants in the monitoring cohort were over 18 months old and at least one year had elapsed since the last dose of sIPV inoculation.Since there is no any data about the protection duration of two-dose Sabin IPV schedules, China CDC propose to follow up the study cohort to evaluate the proportion of seroprotection of antibody and measure neutralizing antibody titers against poliovirus at over 18 months of age infants after a 2-dose or a 3-dose primary schedule of Sabin IPV in Chinese children.

DETAILED DESCRIPTION:
In 2017, China CDC conducted a study titled "A Study of Immunogenicity and Seroconversion With Sabin IPV Schedules in China". This study offers evidence that two doses of sIPV administered at 4 and 8-11 months of age and three doses of sIPV administered at 2, 3, and 4 months of age both provide serological protection against poliomyelitis. At present, all the infants in the monitoring cohort were over 18 months old and at least one year had elapsed since the last dose of sIPV inoculation.

Since there is no any data about the protection duration of two-dose Sabin IPV schedules, China CDC propose to follow up the study cohort when all subjects are at least 18 months old to monitor persistence of antibody. So that, if the antibody levels are not high enough to protect children from the disease, remedial measures can be taken as soon as possible.So China CDC conduct this follow up study ,to

1. Evaluate the proportion of seroprotection of antibody against poliovirus at over 18 months of age infants after a 2-dose or a 3-dose primary schedule of Sabin IPV in Chinese children.
2. Measure neutralizing antibody titers against poliovirus type I, II and III at over 18 months of age infants after 2-dose Sabin IPV schedule, compared with 3-dose Sabin IPV schedule.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian agree to participate in the follow study.
* The subject was vaccinated either two doses or three doses Sabin IPV ,collected two blood samples and laboratory test results were available per protocol of pervious study
* The subject is at least 18 months age.

Exclusion Criteria:

* Parent or legal guardian does not agree to participate in the follow up study.
* The subject has received any polio vaccine product beyond the protocol of previous study.

Ages: 18 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children who had participated the previous Sabin IPV study in 6 counties in Shandong province.
Sampling Method: Non-Probability Sample
Enrollment: 774 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Antibody persistence | 1 month
  Evaluate the proportion of seroprotection of antibody against poliovirus at over 18 months of age infants after a 2-dose or a 3-dose primary schedule of Sabin IPV in Chinese children.

SECONDARY OUTCOMES:
Neutralizing antibody titers | 1 month
  Measure neutralizing antibody titers against poliovirus type I, II and III at over 18 months of age infants after 2-dose Sabin IPV schedule, compared with 3-dose Sabin IPV schedule

CONTACTS AND LOCATIONS:
Overall Officials: Zijian Feng, MD, Study Chair — Centers for Disease Control and Prevention, China; Zhijie An, MPH, Principal Investigator — Centers for Disease Control and Prevention, China; Zundong Yin, Study Director — Centers for Disease Control and Prevention, China
Locations (1):
- Shandong Center for Disease Control and Prevention, Jinan, China

IPD SHARING:
Plan to Share IPD: No